CLINICAL TRIAL: NCT04726384
Title: Physical Activity Level of Patients With COPD During In-hospital Pulmonary Rehabilitation: a Pilot Study
Brief Title: Physical Activity Level of Patients With COPD During Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: OpoleUofTech2
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Physical Activity; SenseWear Armband
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed group: The group was monitored for physical activity levels using the SenseWear Armband device. The group was informed of the purpose of the study and asked to wear the device 24 hours a day for the next 4 days (Friday-Monday) excluding bath time, no more than 30 minutes. Patients received the device on Thursday afternoon and returned it on Tuesday. However, the days Friday-Monday were analyzed to have a record of the entire days
  Interventions: Device: Assessment of physical activity level

INTERVENTIONS:
Device: Assessment of physical activity level — Physical activity was assessed using the Sensewear Armband device. Patients received the device on Thursday mornings, prior to exercise and treatments. The device was placed on the right arm throughout the study. Patients in whom the device monitored a minimum of 95% of the time of the study day were analyzed. Prior to the study, the devices were programmed to record a minimum level of intense (>3MET) and moderate ( >6MET) exercise.

SUMMARY:
The aim of the project was to assess the acceptability of the device as well as adherence to the study. The objective of study was to assess physical activity in patients with COPD during in-hospital pulmonary rehabilitation program. The number of steps, average energy expenditure expressed in MET and kcal, and physical activity time during the consecutive 5 days of the rehabilitation stay were analyzed. Physical activity level was continuously monitored to assess intensity during in-hospital procedures as well as during leisure time.

DETAILED DESCRIPTION:
The aim of the project was to assess the acceptability of the device as well as adherence to the study. The objective of study was to assess physical activity in patients with COPD during in-hospital pulmonary rehabilitation program. The number of steps, average energy expenditure expressed in MET and kcal, and physical activity time during the consecutive 5 days of the rehabilitation stay were analyzed. Physical activity level was continuously monitored to assess intensity during in-hospital procedures as well as during leisure time.

Patients participated in pulmonary rehabilitation program consisted of:

* specific respiratory exercises for 30 minutes - relaxation exercises for breathing muscles, strengthening exercises the diaphragm with resistance, exercises to increase costal or chest breathing, prolonged exhalation exercise, chest percussion, once a day for 30 min,
* training on a cycle ergometer, twice a day for 20-30 min.- until the Heart Rate reaches 70% of the HRmax (220-age),
* fitness exercises - coordination and balance exercises, stretching exercises using elastic bands, balls rehabilitation, sensory pillows. Performed in a standing position, kneeling, sitting, lying on side, abdomen and back, once a day for 30 min
* Schultz autogenic training, once a day 20 min.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD;
* Agreement to participate in the study

Exclusion Criteria:

* Pneumonia, tuberculosis and other respiratory inflammatory disease in all stages and forms
* Condition after a heart attack
* Diabetes
* State after thoracic and cardiac surgery
* Heart failure (stage III, IV ° NYHA)
* Advanced hypertension
* Diseases and injuries that can impair the function of the musculoskeletal system of transportation
* Disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic obstructive pulmonary disease participating in a 3-week hospital-based pulmonary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Energy expenditure - MET | up to 4 days
  The SenseWear Armband was used to assess energy expenditure. The device was used to measure energy expenditure expressed in metabolic equivalent (MET)
Energy expenditure - kcal | up to 4 days
  The SenseWear Armband was used to assess energy expenditure. The device was used to measure energy expenditure expressed in kcal
Number of steps | up to 4 days
  The SenseWear Armband was used to assess number of steps

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Ministry of the Interior and Administration, Głuchołazy, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No